CLINICAL TRIAL: NCT02812927
Title: Study of Glycemic Variability in Post-operative Intensive Care Unit Patients According to Two Insulin Infusion Techniques
Brief Title: Evaluation of Glycemic Variability (GLAIVE)
Acronym: GLAIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2011_17; 2012-A00188-35 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Critical Illness; Anesthesia
Keywords: Glycemic lability index; Continuous glucose monitoring system; intensive care; Insulin
MeSH Terms: conditions — Critical Illness; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard infusion line (Other): The standard insulin infusion system consisted in regular human insulin administration through a six-stopcock manifold connected to the distal line of a multilumen central venous catheter by 150 cm tubing. Insulin was systematically infused by syringe pump on the patient proximal port of the manifold. Carrier was infused via pump through the manifold. All others medicines were infused through the other five stopcocks.
  Interventions: Device: Standard infusion line
- Optimised infusion line (Experimental): The optimised insulin infusion system consisted in regular human insulin administration through a multilumen device (Edelvaiss Multiline-8, Doran International, Toussieu, France). This device had ports for eight infusions which run through separate channels within a 150 cm flexible plastic tube. Since fluids from the individual channels do not meet until they exit the distal tip. Carrier was infused through the high flow (HF) line and insulin was infused by syringe pump systematically next to the HF line port. All others medicines were administered via adjacent ports on the Multiline-8.
  Interventions: Device: Edelvaiss Multiline-8

INTERVENTIONS:
Device: Edelvaiss Multiline-8 — Optimised infusion line
  Arms: Optimised infusion line
Device: Standard infusion line
  Arms: Standard infusion line

SUMMARY:
This study compared two methods of insulin infusion by syringe pumps to assess the impact of medical devices on the glycaemic variability in patients under IIT in ICU. The main objective of the study was to show the superiority of the infusion system which permitted to dedicate a line for the insulin administration on the "standard" installation in terms of control of glycaemic variability.

ELIGIBILITY:
Inclusion Criteria:

* Patients under postoperative intensive care
* Treatment with insulin on bi-lumen central venous catheter over than 48 hours
* Eligibility for interstitial glucose monitoring
* Blood glucose control every 3 hours

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient unwilling to participate in the study
* Patients participating in another study biomedical over the same period
* Patient can not understand the study and its objectives
* Patient under guardianship, curatorship
* Patient malnourished (BMI <18 kg / m²)
* Patient with morbid obesity (BMI> 40 kg / m²)
* Patient in shock (septic or hemodynamic)
* Patients refusing to sign the Medtronic consent on the storage of personal data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2012-09; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
index GLI (Glycemic Lability Index) | up to 48 hours
  This index is calculated from capillary blood glucose.

SECONDARY OUTCOMES:
Number of hypoglycaemic events | 48 hours
  Prevalence and incidence of hypoglycemia
Number of hyperglycaemic events | 48 hours
  Prevalence and incidence of hyperglycemia
Sequential Organ Failure Assessment score (SOFA) | during the 4 days of hospitalization period
  for measure morbidity and mortality
length of stay in Intensive Care Unit (ICU) or in hospital | during the 4 days of hospitalization period
  for measure morbidity and mortality
Death rate | during the 4 days of hospitalization period
  for measure morbidity and mortality
Mean Amplitude Glycemic Excusions score (MAGE) | every 3 hours during 48 hours
  Glycaemic variability
standard deviation of blood glucose | every 3 hours during 48 hours
  Glycaemic variability
average blood glucose | every 3 hours during 48 hours
  Glycaemic variability

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD, PhD, Principal Investigator — University Hospital of Lille

IPD SHARING:
Plan to Share IPD: Undecided